CLINICAL TRIAL: NCT03004300
Title: Maxillary Expansion Effects in the Facial Structures of Children With Upper Airway Obstruction: a Randomized Clinical Trial
Brief Title: Maxillary Expansion Effects in Children With Upper Airway Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, José Valladares Neto, PHD Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 044029
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Airway Obstruction
Keywords: maxillary expansion; adenotonsillar hypertrophy; airway volume
MeSH Terms: conditions — Airway Obstruction | interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Active Comparator): Patients with atresic maxilla without upper airway obstruction submitted to rapid maxillary expansion
  Interventions: Procedure: Rapid maxillary expansion
- group 2 (Experimental): Patients with atresic maxilla and adenotonsillar hypertrophy submitted to rapid maxillary expansion before adenotonsillectomy
  Interventions: Procedure: Rapid maxillary expansion; Procedure: Adenotonsillectomy
- group 3 (Experimental): Patients with atresic maxilla and adenotonsillar hypertrophy submitted to rapid maxillary expansion after adenotonsillectomy
  Interventions: Procedure: Rapid maxillary expansion; Procedure: Adenotonsillectomy

INTERVENTIONS:
Procedure: Rapid maxillary expansion — Device
  Other Names: maxillary expansion
Procedure: Adenotonsillectomy — Surgery
  Arms: group 2; group 3

SUMMARY:
The most frequent causes of mouth breathers are the adenotonsillar hypertrophy. Adenotonsillectomy is the main choice for the elimination of the obstruction. However, this surgical treatment does not have its effect well elucidated and apnea has been cited in the literature as a residual outcome. Other types of supporting treatment may also been involved such as the use of corticosteroids, physiotherapy and orthodontic-orthopedic treatment, among them rapid maxillary expansion (RME).

RME corrects the morphological constriction of the upper arch caused by buccal breathing and also reduce the airway resistance. Despite reports of RME influencing volume enhancement in pharyngeal airway, there are still few three-dimensional studies following the post-expansion effects. In addition, these changes are doubtful due postural changes of the tongue during the tomography exam. Conflicts of results are also present for changes in the nasal septum of children. The main alteration mentioned is the increase in the length of the lower third of the septum.

The investigators propose a randomized, prospective, controlled clinical trial in patients with atresic maxilla with or without adenotonsillar hypertrophy. The patients will be treated with RME and adenotonsillectomy when the obstruction is present. The purpose of this study is elucidate if there is different outcomes considering the moment of RME treatment before or after the adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* Children (boys and girls) between 5 and 9 years of age.
* Atresic maxilla.
* Skeletal Class I
* With or without Adenotonsillar hypertrophy
* Parents or tutors sign Informed Consent.

Exclusion Criteria:

* Craniofacial syndromes or neurologic disease diagnosis.
* History of adenotonsillectomy and orthodontic treatment
* History of facial trauma
* Morbid obesity
* Premature loss of posterior teeth

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Airway Volume | 7 months
  cone beam computed tomography

SECONDARY OUTCOMES:
Quality of life before and after maxillary expansion: | 1 and 7 months
  Obstructive Sleep Apnea-18 questionnaire (OSA-18: scale range 18-126. The impact on quality of life was classified in three groups: a) minor (scores below 60); b) moderate (scores between 60 and 80) and major (scores above 80).
Pediatric Quality of Life | 1 and 7 months
  Pediatric Quality of Life Inventory: 0-100 scale range. Higher scores indicate better HRQOL (Health-Related Quality of Life)
Sleep Disturbance for Children | 1 and 7 months
  Sleep Disturbance Scale for Children: scale range 26-130.Scores higher than 39 indicate sleep disturbance
Nasal septum morphology | 7 months
  Linear parameters by lateral tomographic distances
Dental arch distances | 7 months
  Dental arch growth as described by Mc Namara,2003
Airway obstruction | 7 months
  Adenotonsillar hypertrophy by nasal flexible fiberoptic endoscopy
Bruxism | 7 months
  Bruxism episodes

CONTACTS AND LOCATIONS:
Overall Officials: Jose Valladares Neto, PHD, Principal Investigator — Universidade Federal de Goiás
Locations (1):
- Faculdade de Odontologia, Goiás, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guilleminault C, Monteyrol PJ, Huynh NT, Pirelli P, Quo S, Li K. Adeno-tonsillectomy and rapid maxillary distraction in pre-pubertal children, a pilot study. Sleep Breath. 2011 May;15(2):173-7. doi: 10.1007/s11325-010-0419-3. Epub 2010 Sep 17. PMID 20848317
- [Background] de Castilho LS, Abreu MH, de Oliveira RB, Souza E Silva ME, Resende VL. Factors associated with mouth breathing in children with -developmental -disabilities. Spec Care Dentist. 2016 Mar-Apr;36(2):75-9. doi: 10.1111/scd.12157. Epub 2016 Jan 13. PMID 26763202
- [Background] Caprioglio A, Meneghel M, Fastuca R, Zecca PA, Nucera R, Nosetti L. Rapid maxillary expansion in growing patients: correspondence between 3-dimensional airway changes and polysomnography. Int J Pediatr Otorhinolaryngol. 2014 Jan;78(1):23-7. doi: 10.1016/j.ijporl.2013.10.011. Epub 2013 Oct 25. PMID 24231036
- [Background] Chang Y, Koenig LJ, Pruszynski JE, Bradley TG, Bosio JA, Liu D. Dimensional changes of upper airway after rapid maxillary expansion: a prospective cone-beam computed tomography study. Am J Orthod Dentofacial Orthop. 2013 Apr;143(4):462-70. doi: 10.1016/j.ajodo.2012.11.019. PMID 23561406
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Bruni O, Ottaviano S, Guidetti V, Romoli M, Innocenzi M, Cortesi F, Giannotti F. The Sleep Disturbance Scale for Children (SDSC). Construction and validation of an instrument to evaluate sleep disturbances in childhood and adolescence. J Sleep Res. 1996 Dec;5(4):251-61. doi: 10.1111/j.1365-2869.1996.00251.x. PMID 9065877
- [Background] Fernandes FM, Teles Rda C. Application of the Portuguese version of the Obstructive Sleep Apnea-18 survey to children. Braz J Otorhinolaryngol. 2013 Nov-Dec;79(6):720-6. doi: 10.5935/1808-8694.20130132. PMID 24474484